CLINICAL TRIAL: NCT02466529
Title: Natural History of Spinal Muscular Atrophy Type 1 in Taiwan
Status: Completed | Type: Observational
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Collaborators: Biogen (Industry); Taipei Medical University WanFang Hospital (Other); Taipei Veterans General Hospital, Taiwan (Other Government); Mackay Memorial Hospital (Other); Chang Gung Memorial Hospital (Other); China Medical University Hospital (Other); Chung Shan Medical University (Other); Changhua Christian Hospital (Other); Taichung Veterans General Hospital (Other); Chi Mei Medical Hospital (Other); Cathay General Hospital (Other); Shin Kong Wu Ho-Su Memorial Hospital (Other); Kaohsiung Veterans General Hospital. (Other); National Cheng-Kung University Hospital (Other); Buddhist Tzu Chi General Hospital (Other); Kaohsiung Medical University (Other); Taipei Medical University Shuang Ho Hospital (Other); National Taiwan University Hospital (Other); Taipei Medical University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SMA-NHR10311
Record Dates: First submitted 2015-06-02; First posted 2015-06-09 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-02

CONDITIONS: Natural History of Type 1 Spinal Muscular Atrophy (SMA)
Keywords: type 1 spinal muscular atrophy (SMA)

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- type 1 spinal muscular atrophy: The age of onset of patients with type 1 SMA is below 6 months of age.

SUMMARY:
Spinal muscular atrophy (SMA) is an autosomal recessive disorder characterized by degeneration of motor neurons in the spinal cord and caused by mutations of the survival motor neuron 1 (SMN1) gene.

The investigators will conduct a systematic review of the contents and activities collected via a comprehensive case report form. Patients who fulfilled diagnostic criteria for SMA type 1 will be reviewed retrospectively.

DETAILED DESCRIPTION:
The primary objective of this study is to investigate the natural history of patients with spinal muscular atrophy (SMA) type 1 in Taiwan. This study will provide further insights into the clinical course and pathogenesis of SMA. Several analyses will be conducted regarding overall survival, respiratory support, feeding and nutritional support. The following outcome variables will be examined: correlation between SMA genotype and phenotype, survival, age of onset, and age of confirmed diagnosis, proportion of patients using non-invasive and invasive respiratory support, time to first use of respiratory support, proportion of patients on permanent ventilation, and time to permanent ventilation, number and average duration of hospitalizations, proportion of patients with gastrostomy, number of non-serious and serious respiratory infections, trend of growth parameter (e.g., body weight).

ELIGIBILITY:
Inclusion Criteria:

* Jan. 1979~ 30 Jun. 2014 diagnosed with Spinal Muscular Atrophy (SMA)Type 1
* Onset of paralytic floppy infant less than 6 months of age
* Generalized hypotonia and symmetric weakness, which weakness is more severe in proximal than distal part of extremities
* Weakness in the legs is greater than in the arms
* Tendon reflexes are absent
* Neurogenic changes in electromyogram and/or muscle pathology
* SMN1 gene deletion or mutation

Exclusion Criteria:

* Non-5q SMA (no deletion or mutation of SMN1 gene)
* SMA type 2, type 3 or type 4 (onset of SMA after 6 months of age)

Max Age: 36 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Spinal muscular atrophy Type 1
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2015-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Age of death | up to 36 years
  participants will be followed till the age of death

SECONDARY OUTCOMES:
Age of permanent ventilation | up to 36 years
  participants will be followed till ventilation used 24 hours/day

OTHER OUTCOMES:
Clinical outcome with the following measures-1 | up to 36 years
  Age of onset
Clinical outcome with the following measures-2 | up to 36 years
  Copy numbers of SMN2 gene
Clinical outcome with the following measures-3 | up to 36 years
  Methods of Nutritional Supportive
Clinical outcome with the following measures-4 | up to 36 years
  Methods of Respiratory Supportive

IPD SHARING:
Plan to Share IPD: No